CLINICAL TRIAL: NCT02541695
Title: Characterization Of Resistance Against Live-attenuated Diarrhoeagenic E. Coli
Acronym: CORAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL54064.081.15
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Diarrhea; Gastroenteritis; Bacterial Infections; Escherichia Coli Infections
Keywords: Experimental challenge trial
MeSH Terms: conditions — Diarrhea; Gastroenteritis; Bacterial Infections; Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1E10 CFU Escherichia coli (E. coli) (Active Comparator): 1E10 Colony Forming Units (CFU) Diarrhoeagenic E. coli (strain E1392-75-2A; collection NIZO food research). Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonization Factor Antigen II (CFA/II) and provides 75% protection against challenge with an LT, ST, CFA/II strain.
  At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E10 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A
- 5E10 CFU Escherichia coli (E. coli) (Experimental): 5E10 Colony Forming Units (CFU) Diarrhoeagenic E. coli (strain E1392-75-2A; collection NIZO food research). Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonization Factor Antigen (CFA/II) and provides 75% protection against challenge with an LT, ST, CFA/II strain.
  At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 5E10 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A

INTERVENTIONS:
Biological: E. coli strain E1392-75-2A — At study day 14, after a standardized evening meal and an overnight fast, subjects will receive a single oral dose of the attenuated diarrhoeagenic E. coli strain E1392-75-2A (dose will be either 1E10 CFU (n=22) or 5E10 CFU (n=22)). Oral challenge will occur at 10.00 AM. Under supervision of the project team, subjects will get a NaHCO3 solution (100 ml 2% NaHCO3) to neutralize the gastric acid. After 5 minutes, they get a fruit juice (100 ml) containing the attenuated diarrhoeagenic E. coli strain at the above-mentioned dose. Subjects go home, but are not allowed to drink or eat for 1 hour.
  At study day 35, after a standardized evening meal and an overnight fast, all subjects will receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Other Names: Escherichia coli; E1392-75-2A

SUMMARY:
Although the existing diarrhoeagenic Escherichia coli (E. coli) challenge model is already suitable for dietary interventions in its current form, further characterization of the working-mechanism of the attenuated strain and further optimization of the study design will enable the investigators to better select those ingredients that affect the key pathophysiological processes. The aim of the CORAL study is to further characterize and increase the discriminative power of the diarrhoeagenic E. coli challenge model.

DETAILED DESCRIPTION:
Primary Objective:

In the CORAL study the investigators want to determine whether increasing the inoculation dose of diarrhoeagenic Escherichia coli (E. coli) to 5E10 Colony Forming Units (CFU) (at day 14) and addition of a second challenge 1E10 CFU (at day 35) will result in an increased effect-size and duration of measurable outcomes and in an expansion of the relevant clinical and biomarker readouts of the challenge model.

Secondary Objective:

By extensive biomarker and transcriptome analysis of blood and fecal samples, the investigators aim to explore the working mechanism of the non-toxin producing diarrhoeagenic E. coli strain and the kinetics of the host response to this infection. In addition, the investigators want to determine whether adding extended fasting and addition of a standardized evening meal, prior to the inoculation day, will result in a decreased between-subject variation.

Study design:

The CORAL study is a parallel 7-weeks intervention study. Subjects will be randomly assigned to one of two inoculation dosages of a live attenuated diarrhoeagenic E. coli (n=20 per group). Subjects will be instructed to maintain their usual pattern of physical activity and their habitual food intake, but to standardize their dietary calcium intake. After a standardized evening meal and an overnight fast, subjects will be orally infected with a live, but attenuated, diarrhoeagenic E. coli (strain E1392-75-2A; collection NIZO food research; dose will be either 1E10 CFU (n=22) or 5E10 CFU (n=22) at study day 14). At study day 35, after a standardized evening meal and an overnight fast, all subjects will receive a second inoculation of 1E10 CFU of the ETEC vaccine (n=44).

At various time points before and after both diarrhoeagenic E. coli challenges an online diary will be kept to record all food and drinks consumption to assess dietary macronutrient intake. Moreover, subjects will report information on stool consistency, frequency and severity of symptoms. At various time points before and after both diarrhoeagenic E. coli challenges venous blood and (complete) stool samples will be collected. Blood and fecal samples are collected to quantify several infection- and immune system markers.

Study population:

Healthy male subjects, 18-55 years of age who fulfil all of the inclusion criteria and none of the exclusion criteria will participate in the CORAL study.

Intervention:

At study day 14 and 35, after a standardized evening meal and an overnight fast, all subjects will receive an inoculation of the diarrhoeagenic E. coli (1E10 CFU (n=22) or 5E10 CFU (n=22) at study day 14; 1E10 CFU (n=40) at study day 35) Subjects will be instructed to maintain their habitual diet, except for their dairy intake. Dairy has a high calcium content and contributes significantly to total daily calcium intake. These dietary guidelines will limit calcium intake on average to 500 mg/day. From our previous studies, we know that calcium can significantly reduce the gastro-intestinal symptoms induced by the E. coli strain.

Main study parameter:

1. Percentage of faecal dry weight (% determined by freeze-drying)

Secondary study parameters:

1. Total faecal wet weight (faecal weight in g/day)
2. Time to first diarrhoeal stool (reported by the subjects in the online diary)
3. Stool consistency (Bristol Stool Scale reported by the subjects in the online diary
4. Number of stools with Bristol Stool Scale >4 (Bristol Stool Scale reported by the subjects in the online diary)
5. Stool frequency (Stools per day reported by the subjects in the online diary)
6. Incidence and duration of WHO-defined diarrhoea (Calculated from the Bristol Stool Scale and the Stool frequency reported by the subjects in the online diary)
7. The incidence, duration and severity of Gastro-intestinal symptoms (Gastro-intestinal Symptom Rating Scale reported by the subjects in the online diary).
8. In addition, the study contains an explorative phase consisting of biomarker and transcriptome analysis, in order to further explore and identify the mechanism and kinetics of the host response to the infection.

ELIGIBILITY:
Inclusion criteria:

1. Ability to follow verbal and written instructions;
2. Age between 18 and 55 years;
3. Availability of internet connection;
4. BMI ≥20 and ≤27 kg/m2;
5. Healthy as assessed by the NIZO food research medical questionnaire;
6. Male subjects;
7. Signed informed consent;
8. Voluntary participation;
9. Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned;
10. Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years;
11. Willing to comply with study procedures;
12. Willingness to abstain from high calcium containing products.
13. Willingness to abstain from medications that contain acetaminophen, aspirin, ibuprofen, and other nonsteroidal anti-inflammatory drugs, (OTC) antacids and antimotility agents (eg, loperamide) on the three days before, during and 3 days after diarrhoeagenic E. coli challenge.
14. Willingness to abstain from alcoholic beverages three days before, during and three days after diarrhoeagenic E. coli challenge.
15. Willingness to give up blood donation starting 1 month prior to study start and during the entire study;

Exclusion criteria:

1. Disease of the GI tract, liver, bile bladder, kidney, thyroid gland (self-reported);
2. Diarrhoeagenic E.coli strain (as used in the study) detected in fecal sample at screening;
3. Evidence of current excessive alcohol consumption or non-therapeutic drug (ab)use);
4. Evidence of IgA deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay).
5. High titer serum antibodies against CFA-II diarrhoeagenic E.coli strain (as used in the study) at screening;
6. History of microbiologically confirmed ETEC or cholera infection in last 3 years.
7. Known allergy to the following antibiotics: ciprofloxacin, trimethoprim-sulfamethoxazole, and penicillins.
8. Mental status that is incompatible with the proper conduct of the study;
9. Not having a general practitioner, not allowing disclosure of participation to the general practitioner or not allow to inform the general practitioner about abnormal results.
10. Occupation involving handling of ETEC or Vibrio cholerae currently, or in the past 3 years.
11. Participation in any clinical trial including blood sampling and/or administration of substances starting 1 month prior to study start and during the entire study;
12. Personnel of NIZO food research, their partner and their first and second degree relatives;
13. Reported average stool frequency of <1 or >3 per day;
14. Symptoms consistent with Travelers' Diarrhoea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study.
15. Use of antibiotics, norit, laxatives (up till 6 months prior to inclusion), cholestyramine, antacids H2 receptor antagonists or proton pump inhibitors or immune suppressive agents (up till 3 months prior to inclusion);
16. Vaccination for or ingestion of ETEC, cholera, or E coli heat labile toxin within 3 years prior to inclusion;
17. Vegetarians and vegans

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in percentage of faecal dry weight from baseline | Day 14-17 and Day 35-38
  % of faecal dry weight determined by freeze-drying

SECONDARY OUTCOMES:
Change in total faecal wet weight from baseline | Day 14-17 and Day 35-38
  Total faecal weight in g/day
Time to first diarrhoeal stool | Day 14-15 and Day 35-36
  Time to first diarrhoeal stool reported by subjects
Change in Stool frequency from baseline | Day 14-17 and Day 35-38
  Stools per day reported the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Sandra TenBruggencate, PhD, Principal Investigator — NIZO Food Research; Els VanHoffen, PhD, Principal Investigator — NIZO Food Research; Alwine Kardinaal, PhD, Principal Investigator — NIZO Food Research
Locations (2):
- Netherlands (2):
  - NIZO food research, Ede, Gelderland
  - Hospital Gelderse Vallei, Ede, Gelderland

REFERENCES:
- [Background] Bovee-Oudenhoven IM, Lettink-Wissink ML, Van Doesburg W, Witteman BJ, Van Der Meer R. Diarrhea caused by enterotoxigenic Escherichia coli infection of humans is inhibited by dietary calcium. Gastroenterology. 2003 Aug;125(2):469-76. doi: 10.1016/s0016-5085(03)00884-9. PMID 12891550
- [Background] Ouwehand AC, ten Bruggencate SJ, Schonewille AJ, Alhoniemi E, Forssten SD, Bovee-Oudenhoven IM. Lactobacillus acidophilus supplementation in human subjects and their resistance to enterotoxigenic Escherichia coli infection. Br J Nutr. 2014 Feb;111(3):465-73. doi: 10.1017/S0007114513002547. Epub 2013 Aug 12. PMID 23930950
- [Background] Ten Bruggencate SJ, Girard SA, Floris-Vollenbroek EG, Bhardwaj R, Tompkins TA. The effect of a multi-strain probiotic on the resistance toward Escherichia coli challenge in a randomized, placebo-controlled, double-blind intervention study. Eur J Clin Nutr. 2015 Mar;69(3):385-91. doi: 10.1038/ejcn.2014.238. Epub 2014 Nov 5. PMID 25369827
- [Derived] van Hoffen E, Mercenier A, Vidal K, Benyacoub J, Schloesser J, Kardinaal A, Lucas-van de Bos E, van Alen I, Roggero I, Duintjer K, Berendts A, Albers R, Kleerebezem M, Ten Bruggencate S. Characterization of the pathophysiological determinants of diarrheagenic Escherichia coli infection using a challenge model in healthy adults. Sci Rep. 2021 Mar 15;11(1):6060. doi: 10.1038/s41598-021-85161-1. PMID 33723346
- See also: Study location — http://www.nizo.com